CLINICAL TRIAL: NCT04363073
Title: Assessment of Annabella Breast Pump Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Annabella Tech Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: Annabella V1
Record Dates: First submitted 2020-04-17; First posted 2020-04-27 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Breast Feeding
Keywords: Breast Feeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anaabella (Experimental): Milk will be expressed using Annabella breast pump.
  Interventions: Device: Annabella Breast Pump
- Control pump (Active Comparator): Milk will be expressed using a control breast pump.
  Interventions: Device: Control Breast Pump

INTERVENTIONS:
Device: Annabella Breast Pump — Milk will be expressed using Annabella breast pump for 4 consecutive days (at least 24h apart)
  Arms: Anaabella
Device: Control Breast Pump — Milk will be expressed using Control breast pump for 4 consecutive days (at least 24h apart)
  Arms: Control pump

SUMMARY:
This is an interventional, prospective, randomized, comparative, two-period cross over study to evaluate the performance of Annabella breast pump against a control breast pump.

DETAILED DESCRIPTION:
50 women who are 2-5 months post-delivery will be included in the study following appropriate consent. Women will be randomly allocated to two groups for the type of pump used on the first session. Each expression visit will start approximately 3 hours after the end of a regular baby feeding session. Each expression visit will start approximately 3 hours after the end of a regular baby feeding session. During each visit, milk will be expressed once a day from each of the two breasts (left & right). During the 4 first visits (at least 1 day apart) Annabella or the control pump will be used. After at least 3 days washout period, milk will be expressed for additional 4 days, once a day from each of the two breasts, using the other breast pump. An expression session will last until no milk is expressed for 3 min continuously but not for longer than 25 min. Participants will be serving as their own control. Milk will be collected for volume and quality assessment. Maternal comfort at the end of each visit will be assessed using questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Women ≥ 18 years old
* Women whom are 2-5 months post delivery
* Lactating women - Breastfeed with no more than formula feeding twice a day and no solid food feeding (which replace breastfeeding) during the study period.
* Breastfeed or pumping at least 5 times a day
* Mother to healthy infant born at ≥ 37 weeks of gestation age.

Exclusion Criteria:

* Woman who consumes under 1,500 kcal/day (on a diet)
* Report a high mental stress condition and/or depression
* Use of estrogen oral contraceptives
* Pregnant women
* Suffer from chronic diseases that can impact breast feeding
* Participate in another clinical trial
* Mothers of babies who may develop feeding difficulties according to the investigator decisions (such as cleft pallet, autism).
* Woman with Sunken/ flat nipple or inverted nipple. or any other physiological condition that may disturb breast feeding.
* Woman that declares at time of recruitment that she is unable to extract more than 25ml per breastfeeding (overall from both breast)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2020-12-30 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Milk Volume collected using the breast pump | immediately after the intervention
  Total milk Volume (cc)

SECONDARY OUTCOMES:
Satisfaction Satisfaction questionnaires | immediately after the intervention
  rating scale: Min: 1 , Max: 10; higher score- better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Revital Sheinberg, MD, Principal Investigator — Shiba Medical Center, Israel
Locations (1):
- Shamir medical center, Be’er Ya‘aqov, Israel

IPD SHARING:
Plan to Share IPD: No